CLINICAL TRIAL: NCT03837925
Title: Pharmaco-metabolomic Effects of Statins: METASTATINE
Acronym: METASTATINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Fondation Coeur et Recherche (Unknown); ICAN Nutrition Education and Research (Industry); Fédération francaise de cardiologie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-02
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Diseases
Keywords: Statins; cardiovascular risk; primary prevention microbiota; metabolomics
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: 2 groups of patients having treatment or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo manufactured as the treatment. Packaging identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATORVASTATIN (Experimental): Atorvastatin 40mg caps: one daily. 3 patient visits: inclusion / week 2 / week 6. At each visit, blood sampling, stool sampling, ECG, to evaluate the pharmaco-metabolomic effects of the Statine
  Interventions: Drug: Atorvastatin 40mg Tablet
- PLACEBO (Placebo Comparator): Placebo caps: one daily. 3 patient visits: inclusion / week 2 / week 6. At each visit, blood sampling, stool sampling, ECG to compare the pharmaco-metabolomic effects of the Statine between atorvastatin arm and placebo arm
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Atorvastatin 40mg Tablet — Patient participation for 6 weeks of treatment
  Other Names: No other name
  Arms: ATORVASTATIN
Drug: Placebo comparator — Patient participation for 6 weeks of treatment
  Other Names: No other name
  Arms: PLACEBO

SUMMARY:
Statins are effective in cardio-vascular prevention by lowering LDL-Cholesterol levels but also through other mechanisms poorly understood. Our hypothesis is that some of these effects are mediated by microbiota alteration, leading to diminution of expression of microbiota derived pro-atherogenic metabolites.

DETAILED DESCRIPTION:
The aim of this prospective double blind placebo-controlled study is to evaluate the acute effects of statins on microbiota and its derived metabolites at 2 and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cardiovascular risk requiring statins in primary prevention
* Contraception for women of childbearing age

Exclusion Criteria:

* Previous antibiotics, proton pomp inhibitors, statins or other hypolipidemic drugs intake in the previous three months
* Renal insufficiency with creatinine clearance <40ml/min
* Contra-indication to statins
* Previously known conditions affecting muscles, or digestive system
* Requirement of statins in secondary prevention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Rate of trimethylamine N-oxide trimethylamine oxide in blood, measured post-prandially at week-6 in atorvastatin arm and placebo arm. | Week-6
  The main objective of the study is to measure the direct effect of Hydroxy-methyl-glutaryl-coenzyme A reductase inhibitors (Atorvastatin) on the production of atherogenic metabolites derived from intestinal microbiota

SECONDARY OUTCOMES:
Rate of trimethylamine N-oxide trimethylamine oxide in blood, measured post-prandially at week-2 in atorvastatin arm and placebo arm. | week-2
  To evaluate the evolution of the whole circulating metabolomic profile linked to the introduction of statins
Rate of trimethylamine N-oxide trimethylamine oxide in blood, measured pre and post-prandially at week-2 and week-6 in atorvastatin arm. | Week-2 and week-6
  To evaluate changes in the microbiome related to the introduction of statins
Comparison between W0, W2 and W6 after initiation of atorvastatin vs placebo of circulating metabolomic profile (pre- and postprandial) | Week 2 and Week 6
  To correlate changes in lipid parameters induced by statins with metabolomic and lipidemic changes and microbiome. Rate of 100 metabolites will be analysed, and gathered as follows:
  metabolism of acylcarnitine (3), metabolism of bile acids (5), carbohydrate metabolism (1), dietary choline metabolism (3), metabolism of amino acids (34), vitamins and cofactors (7), metabolism of creatine (2), polyamine metabolism (3), purine metabolism (5), pyrimidine metabolism (9), tryptophan / kynurenine metabolism (21), caffeine metabolism (3), Citric Acid cycle (3), urea cycle (1)
Comparison between W0, W2 and W6 after initiation of atorvastatin vs placebo of the microbiome | Week 2 and Week 6
  To analyze the influence of the microbiota on the variability of response to atorvastatin.
  169/5000 The stool will be analyzed by metagenomic sequencing using the "shot gun" technique, a direct sequencing that quantifies the number of bacterial genes and annotates them.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Elie SALEM, MD, Principal Investigator — CIC 1421 CHU Pitie Salpetriere
Locations (2):
- France (2):
  - CIC La Sapétrière, Paris
  - CIC HEGP, Paris

IPD SHARING:
Plan to Share IPD: No